CLINICAL TRIAL: NCT02707068
Title: Quality Of LIfe Tool for IBD (QOLITI): Pilot Testing of a Self-administered Intervention to Target Psychological Distress in Inflammatory Bowel Disease
Brief Title: Quality Of LIfe Tool for IBD
Acronym: QOLITI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RJ116/N006
Record Dates: First submitted 2016-02-04; First posted 2016-03-14 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2016-04

CONDITIONS: Inflammatory Bowel Disease
Keywords: Quality of Life; Self-help intervention
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- QOLITI (Experimental): Intervention group receives the QOLITI ("Quality Of LIfe Tool for IBD") manual immediately to work with over the course of several weeks along with 3 x 30 minutes of telephone support by a trained healthcare professional. Telephone calls will occur at two, four and six weeks post-randomisation.
  Participants will be invited to discuss their experiences after the end of the actual study. These interviews are no obligatory part of the QOLITI study.
  Interventions: Behavioral: Quality Of LIfe Tool for IBD (QOLITI)
- Waitlist Control group (WLC) (No Intervention): Waitlist control group waits until after the study finishes to receive the same manual, but without telephone support sessions.

INTERVENTIONS:
Behavioral: Quality Of LIfe Tool for IBD (QOLITI) — The cognitive-behavioural therapy (CBT)-inspired manual will contain several chapters each of which addresses a different topic with information, guidance in setting goals for behaviour change and accompanying tasks to aid implementation which will be completed at home in the participant's own time. Key themes are likely to include symptom management, dealing with social implications of the disease and interacting effectively with healthcare professionals among others. Each chapter will address a theme providing information, sign posting to appropriate organisations, step-by-step tasks and quotes from pwIBD among others, drawing on relevant therapeutic approaches for self-management including CBT and certain elements of Acceptance and Commitment Therapy.
  Arms: QOLITI

SUMMARY:
This study seeks to test the feasibility of a self-management manual with minimal telephone support by a healthcare professional. The study will also explore the acceptability of the intervention manual to patients.

DETAILED DESCRIPTION:
Psychological distress and poor quality of life are common in Long Term Conditions (LTCs) including Inflammatory Bowel Disease (IBD). Rates of depression are 11-21% in people with IBD (pwIBD) with high levels of anxiety in 41%. Additionally, as diagnosis typically occurs at 15-40 years, educational and employment attainment can be effected and symptoms and medical procedures such as diarrhoea and colonoscopies can be stressful and embarrassing. The relapsing and remitting nature can also cause uncertainty and fear of social integration.

Most of the psychosocial literature in IBD has focused on the potential impact of stress and recording the prevalence and non-modifiable predictors of depression and anxiety such as active disease, hospitalisation, surgery (particularly stoma formation) and unemployment. Less research in IBD has investigated potentially modifiable factors known to be related to distress and quality of life in other LTCs such as illness perceptions, social support and coping strategies, although one study has found a similar association in IBD. This is of particular interest due to the potential behavioural and physiological pathways through which they could impact on health and quality of life.

Psychosocial interventions in IBD to date have focused on stress management or Cognitive Behavioural Therapy (CBT) to reduce distress and improve quality of life. Although small sample studies have shown small to moderate benefits of the interventions, these approaches are time consuming and resource intensive such as group or individual therapy. This can result in low adherence and retention due to the required time commitment, but more importantly are not widely applicable in the NHS due to limited available expertise and in particular, their cost. Psychological interventions are most effective when tailored specifically to disease-related factors and the patients' developmental stage. Such interventions are currently lacking for IBD.

An alternative to therapist-led intervention is to promote self-management through paper or online self-help interventions supplemented by minimal guided support by a health care professional. This type of supported, self-directed intervention is cost-effective and has shown strongest results when targeted to the needs of specific diseases. There is currently no similar self-directed manual for IBD available. This type of supported, self-directed intervention can be incorporated into standard care where required, is cost-effective and has the potential to support pwIBD to successfully adjust to their LTC for better clinical and quality of life outcomes. Although most people will not require intensive psychological therapy for debilitating distress, structured support to adjust to the many demands that IBD places on people could help to bridge the gap for the 40-50% of pwIBD that show moderate levels of distress, improving their quality of life and management of the illness.

Sample size justification: A sample size of 30 per group is in line with recommendations for pilot studies where the aim is to determine the feasibility of a future efficacy study by estimating the treatment effect (for a power calculation) and estimating rate of non-completion of the intervention. A minimum total sample size of 50 (i.e. 25 per group) is recommended to allow for a precise estimate of the pooled standard deviation at the post intervention assessment. Increasing the number to 30 per group allows for non-completion of up to 20%. Furthermore, a sample size of 30 per group allows for an acceptably precise estimate of the non-completion rate; a 95% confidence interval less than +/-11% for completion rates of 80% or higher.

Adults (>18 years) with IBD will be provided with an information sheet and invited to participate in the study. Following informed consent and the completion of baseline questionnaires, participants will be randomised to receive either intervention + treatment as usual (treatment group) or treatment as usual (control group). Randomisation will be completed by King's College London Clinical Trials Unit independently of the research team so that the researchers remain blind to condition.

As recommended for a pilot or feasibility study, results will be mainly descriptive and will include; proportion of eligible people; consent rate; retention rate. The investigators plan on using an intention-to-treat regression analysis and include the pre measure as a covariate. This data will allow for effect sizes and feasibility to be determined in order to adequately power a full trial of the intervention in a follow-up study. Thematic analysis of the qualitative feedback data will be conducted by a member independent of the research team.

ELIGIBILITY:
Inclusion Criteria:

* Participants with must have a diagnosis of IBD,
* be over 18 years of age as well as able to read and understand English fluently.
* Informed consent must be obtained.

Exclusion Criteria:

* Participants are not eligible for the study, if they do not fulfil the inclusion criteria.
* Suicidal patients will be directly referred to liaison psychiatry or their GP and will not be able to access the study as the intensity of the manual intervention is within the low-moderate range and thus not suitable to address severe symptoms appropriately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Feasibility | within 2 weeks of potential participants getting in touch (i.e. once at the beginning of the study)
  Percentage of patients eligible
Acceptability | within 2 weeks of potential participants getting in touch (i.e. once at the beginning of the study)
  Percentage of eligible patients consenting
Effectiveness: Change in depression | within 2 weeks of obtaining consent as well as 10 weeks post-randomisation
  Assessing whether depression levels have changed from pre- to post-intervention (Patient Health Questionnaire, PHQ-9)
Acceptability: Change in numbers of participants throughout the trial | 2 weeks of obtaining consent compared to 10 weeks post-randomisation
  Percentage of consenting eligible participants retained until completion
Effectiveness: Change in anxiety | within 2 weeks of obtaining consent as well as 10 weeks post-randomisation
  Assessing whether anxiety levels have changed from pre- to post-intervention (Generalised Anxiety Disorder 7-item scale, GAD-7)
Effectiveness: Change in generic quality of life | within 2 weeks of obtaining consent as well as 10 weeks post-randomisation
  Assessing whether generic quality of life levels have changed from pre- to post-intervention (EQ-5D-5L)
Effectiveness: Change in Inflammatory Bowel Disease - specific quality of life | within 2 weeks of obtaining consent as well as 10 weeks post-randomisation
  Assessing whether IBD-specific quality of life levels have changed from pre- to post-intervention (Inflammatory Bowel Disease Questionnaire, IBDQ)

SECONDARY OUTCOMES:
Semi-structured qualitative interviews | at 12 weeks post-randomisation
  semi-structured qualitative interviews of up to 30 minutes to obtain retrospective appraisal of the intervention (i.e. content and layout), conducted by a person independent of the research group, transcribed data will be analysed based on principles of grounded theory
Change in fatigue | within 2 weeks of obtaining consent as well as 10 weeks post-randomisation
  Assessing whether fatigue levels have changed from pre- to post-intervention (Chalder Fatigue Scale, CFS)
Change in illness perception | within 2 weeks of obtaining consent as well as 10 weeks post-randomisation
  Assessing whether illness perception has changed from pre- to post-intervention (Illness Perception Questionnaire, IPQ-R)
Change in disease activity | within 2 weeks of obtaining consent as well as 10 weeks post-randomisation
  Assessing whether subjective levels if disease activity have changed from pre- to post-intervention (patient-modified Simple Clinical Colitis Activity Index, p-SCCAI)
Change in disease activity | within 2 weeks of obtaining consent as well as 10 weeks post-randomisation
  Assessing whether subjective levels if disease activity have changed from pre- to post-intervention (Crohn's Disease Activity Index for research surveys, CDAI for research surveys)

CONTACTS AND LOCATIONS:
Overall Officials: Lynsady D Hughes, PhD, Principal Investigator — King's College London
Locations (1):
- Health Psychology Section, Psychology Dept, Institute of Psychiatry, King's College London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The investigators seek to publish the results of the study which are going to be based on group statistics only, i.e. no individual patient data will be made available.

REFERENCES:
- [Background] Graff LA, Walker JR, Clara I, Lix L, Miller N, Rogala L, Rawsthorne P, Bernstein CN. Stress coping, distress, and health perceptions in inflammatory bowel disease and community controls. Am J Gastroenterol. 2009 Dec;104(12):2959-69. doi: 10.1038/ajg.2009.529. Epub 2009 Sep 15. PMID 19755973
- [Background] Tang LY, Nabalamba A, Graff LA, Bernstein CN. A comparison of self-perceived health status in inflammatory bowel disease and irritable bowel syndrome patients from a Canadian national population survey. Can J Gastroenterol. 2008 May;22(5):475-83. doi: 10.1155/2008/109218. PMID 18478133
- [Background] Nahon S, Lahmek P, Durance C, Olympie A, Lesgourgues B, Colombel JF, Gendre JP. Risk factors of anxiety and depression in inflammatory bowel disease. Inflamm Bowel Dis. 2012 Nov;18(11):2086-91. doi: 10.1002/ibd.22888. Epub 2012 Jan 31. PMID 22294486
- [Background] Huppe A, Langbrandtner J, Raspe H. [Assessing complex health problems of patients with IBD--first step to patient activation]. Z Gastroenterol. 2013 Mar;51(3):257-70. doi: 10.1055/s-0032-1325354. Epub 2013 Mar 13. German. PMID 23487355
- [Background] Marri SR, Buchman AL. The education and employment status of patients with inflammatory bowel diseases. Inflamm Bowel Dis. 2005 Feb;11(2):171-7. doi: 10.1097/00054725-200502000-00011. PMID 15677911
- [Background] Denters MJ, Schreuder M, Depla AC, Mallant-Hent RC, van Kouwen MC, Deutekom M, Bossuyt PM, Fockens P, Dekker E. Patients' perception of colonoscopy: patients with inflammatory bowel disease and irritable bowel syndrome experience the largest burden. Eur J Gastroenterol Hepatol. 2013 Aug;25(8):964-72. doi: 10.1097/MEG.0b013e328361dcd3. PMID 23660935
- [Background] Moradkhani A, Beckman LJ, Tabibian JH. Health-related quality of life in inflammatory bowel disease: psychosocial, clinical, socioeconomic, and demographic predictors. J Crohns Colitis. 2013 Jul;7(6):467-73. doi: 10.1016/j.crohns.2012.07.012. Epub 2012 Aug 10. PMID 22884758
- [Background] Triantafillidis JK, Merikas E, Gikas A. Psychological factors and stress in inflammatory bowel disease. Expert Rev Gastroenterol Hepatol. 2013 Mar;7(3):225-38. doi: 10.1586/egh.13.4. PMID 23445232
- [Background] Bonaz BL, Bernstein CN. Brain-gut interactions in inflammatory bowel disease. Gastroenterology. 2013 Jan;144(1):36-49. doi: 10.1053/j.gastro.2012.10.003. Epub 2012 Oct 12. PMID 23063970
- [Background] Knowles SR, Cook SI, Tribbick D. Relationship between health status, illness perceptions, coping strategies and psychological morbidity: a preliminary study with IBD stoma patients. J Crohns Colitis. 2013 Nov;7(10):e471-8. doi: 10.1016/j.crohns.2013.02.022. Epub 2013 Mar 28. PMID 23541738
- [Background] Keefer L, Doerfler B, Artz C. Optimizing management of Crohn's disease within a project management framework: results of a pilot study. Inflamm Bowel Dis. 2012 Feb;18(2):254-60. doi: 10.1002/ibd.21679. Epub 2011 Feb 23. PMID 21351218
- [Background] Thompson RD, Craig A, Crawford EA, Fairclough D, Gonzalez-Heydrich J, Bousvaros A, Noll RB, DeMaso DR, Szigethy E. Longitudinal results of cognitive behavioral treatment for youths with inflammatory bowel disease and depressive symptoms. J Clin Psychol Med Settings. 2012 Sep;19(3):329-37. doi: 10.1007/s10880-012-9301-8. PMID 22699797
- [Background] Taylor RS, Watt A, Dalal HM, Evans PH, Campbell JL, Read KL, Mourant AJ, Wingham J, Thompson DR, Pereira Gray DJ. Home-based cardiac rehabilitation versus hospital-based rehabilitation: a cost effectiveness analysis. Int J Cardiol. 2007 Jul 10;119(2):196-201. doi: 10.1016/j.ijcard.2006.07.218. Epub 2006 Nov 7. PMID 17084927
- [Background] van Kessel K, Moss-Morris R, Willoughby E, Chalder T, Johnson MH, Robinson E. A randomized controlled trial of cognitive behavior therapy for multiple sclerosis fatigue. Psychosom Med. 2008 Feb;70(2):205-13. doi: 10.1097/PSY.0b013e3181643065. Epub 2008 Feb 6. PMID 18256342
- [Background] Moss-Morris R, McAlpine L, Didsbury LP, Spence MJ. A randomized controlled trial of a cognitive behavioural therapy-based self-management intervention for irritable bowel syndrome in primary care. Psychol Med. 2010 Jan;40(1):85-94. doi: 10.1017/S0033291709990195. Epub 2009 Jun 17. PMID 19531276
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Cheung WY, Garratt AM, Russell IT, Williams JG. The UK IBDQ-a British version of the inflammatory bowel disease questionnaire. development and validation. J Clin Epidemiol. 2000 Mar 1;53(3):297-306. doi: 10.1016/s0895-4356(99)00152-3. PMID 10760641
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391